CLINICAL TRIAL: NCT01155167
Title: The Effect of Topical Administration of Lidocaine/Nitroglycerin Combination Versus Placebo on Radial Artery Access in Patients Undergoing Cardiac Catheterization Via the Radial Artery
Brief Title: Topical Radial Artery Vasodilation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10035824; CHR # 10035824 (Other: UCSF)
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Results first posted 2013-05-15 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2013-05

CONDITIONS: Cardiac Catheterization; Spasm
Keywords: radial artery spasm
MeSH Terms: conditions — Spasm | interventions — Nitroglycerin; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Topical dilator (Experimental)
  Interventions: Drug: Nitroglycerin and lidocaine

INTERVENTIONS:
Drug: Nitroglycerin and lidocaine — Topical Nitroglycerin and lidocaine
  Arms: Topical dilator
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of the study is to facilitate radial artery access for cardiac catheterization. The investigators hypothesize that topical nitroglycerin and lidocaine will reduce radial artery spasm. Patients undergoing cardiac catheterization via the radial artery will be randomized to topical nitroglycerin + lidocaine versus placebo.

DETAILED DESCRIPTION:
The aim of the study is to facilitate radial artery access for cardiac catheterization. The investigators hypothesize that topical nitroglycerin and lidocaine will reduce radial artery spasm. Patients undergoing cardiac catheterization via the radial artery will be randomized to topical nitroglycerin + lidocaine versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing trans-radial cardiac catheterization

Exclusion Criteria:

* inability to receive nitroglycerin or lidocaine due to allergy or medication interactions

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Boyle, MBBS, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco Medical Center, San Francisco, California, United States

REFERENCES:
- [Derived] Beyer AT, Ng R, Singh A, Zimmet J, Shunk K, Yeghiazarians Y, Ports TA, Boyle AJ. Topical nitroglycerin and lidocaine to dilate the radial artery prior to transradial cardiac catheterization: a randomized, placebo-controlled, double-blind clinical trial: the PRE-DILATE Study. Int J Cardiol. 2013 Oct 3;168(3):2575-8. doi: 10.1016/j.ijcard.2013.03.048. Epub 2013 Apr 10. PMID 23582415

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients scheduled to undergo clinically indicated diagnostic or therapeutic cardiac catheterization via the transradial approach were invited to participate in the study
Pre-assignment Details: 3 participants from the placebo group were excluded (2 secondary to insufficient or uninterpretable ultrasound data and 1 secondary to patient's access site change from transradial access (TRA) to femoral access).
Groups:
- Placebo: Two placebo topical lotions (chosen to resemble the appearance of the active creams) were applied to the radial artery site and covered by transparent film dressing for at least 30 minutes prior to the radial artery access time.
- Topical Dilator: 40mg of lidocaine cream + 30mg nitroglycerin ointment were applied to the radial artery site and covered by transparent film dressing for at least 30 minutes prior to the radial artery access time.
Period: Overall Study
Arm/Group | Placebo | Topical Dilator
Started | 43 | 43
Completed | 40 | 43
Not Completed | 3 | 0
Not completed — Insufficient ultrasound data | 2 | 0
Not completed — Access site changed to femoral artery | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Two topical placebo lotions (chosen to resemble the appearance of the active creams) were applied to the radial artery site and covered by transparent film dressing for at least 30 minutes prior to the radial artery access time.
- Total: Total of all reporting groups
Arm/Group | Placebo | Topical Dilator | Total
Number analyzed (Participants) | 40 | 43 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 22 | 43
  >=65 years | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (12.8) | 63.4 (12.6) | 61.2 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 26 | 29 | 55
Region of Enrollment [Number; unit: participants]
  United States | 40 | 43 | 83

OUTCOME MEASURES:

1. Primary Outcome: Change in Radial Artery Diameter
Description: The cross-sectional radial artery area was measured using a high frequency linear array transducer. All ultrasound measurements were made 2 cm proximal to the radial styloid process. Each measurement was performed 3 times and averaged. At least 30 minutes after the application of topical creams, the radial artery diameter was again measured in the same fashion.
Time Frame: Baseline and after 30 minutes of drug application
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Topical Dilator
Number analyzed (Participants) | 40 | 43
Percent change | -5.6 (2.1) | 16.5 (4.2)

2. Secondary Outcome: Radial Artery Spasm During Catheterization
Description: The blinded clinical operator recorded whether radial artery spasm occurred, as detected by resistance to advancing the catheter through the radial artery, by difficulty in torquing the catheter, or by difficulty in removing the catheter.
Time Frame: 2 hours
Population: All participants except 3 participants in the Topical Dilator arm for whom RAS data were not recorded
Measure: Number; unit: participants
Arm/Group | Placebo | Topical Dilator
Number analyzed (Participants) | 40 | 40
participants
  Spasm | 10 | 10
  No spasm | 30 | 30

3. Secondary Outcome: Radial Artery Patency
Description: Prior to discharge, color doppler ultrasound was used at the site where the sheath had been inserted to determine whether the radial artery was patent (open, unobstructed).
Time Frame: 24 hours
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Placebo | Topical Dilator
Number analyzed (Participants) | 40 | 43
participants
  Patent radial artery | 39 | 43
  Early radial artery occlusion | 1 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Topical Dilator
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/40 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No